CLINICAL TRIAL: NCT04838847
Title: COVID-19 (CoviCompareCV): A Phase 3, Non-randomized, Open Label Clinical Trial to Evaluate the Immunogenicity and Safety of the Investigational SARS-CoV-2 mRNA Vaccine CVnCoV Administered Intramuscularly in Adults Aged 65 Years or Above Compared to Younger Adults Aged 18-45 Years
Brief Title: A Study to Evaluate the Immunogenicity and Safety of the SARS-CoV-2 mRNA Vaccine CVnCoV in Elderly Adults Compared to Younger Adults for COVID-19
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was withdrawn based on an assessment of immunogenicity in elderly adults.
Sponsor: CureVac (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CV-NCOV-012; 2020-005064-54 (EudraCT Number)
Record Dates: First submitted 2021-04-08; First posted 2021-04-09 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-04

CONDITIONS: Coronavirus; Covid19; SARS-CoV-2; Severe Acute Respiratory Syndrome
Keywords: Covid19; SARS-CoV-2 mRNA vaccine; CVnCoV; Vaccine; SARS; COVID; Safety; Immunogenicity
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Severe Acute Respiratory Syndrome | interventions — CVnCoV COVID-19 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants / Healthy Participants Aged ≥65 Years (Experimental): Participants will be vaccinated with CVnCoV 12 μg mRNA on Day 1 and Day 29 in the deltoid area, preferably in the non-dominant arm.
  Interventions: Biological: CVnCoV Vaccine
- Participants / Healthy Participants Aged 18-45 Years (Experimental): Participants will be vaccinated with CVnCoV 12 μg mRNA on Day 1 and Day 29 in the deltoid area, preferably in the non-dominant arm.
  Interventions: Biological: CVnCoV Vaccine

INTERVENTIONS:
Biological: CVnCoV Vaccine — Intramuscular (IM) injection
  Other Names: CV07050101

SUMMARY:
The primary objective of this study is to evaluate the humoral immune response to CVnCoV in elderly adults aged ≥65 years and younger adults aged 18-45 years, 14 days after the second dose administration.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants between the ages of 18 and 45 years or aged 65 years and older.
2. Healthy adults or adults with pre-existing medical conditions who are in a stable condition. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during 3 months before enrollment.
3. Capable of giving personal signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form and in this study protocol.
4. Physical examination without clinically significant findings according to the Investigator's assessment.
5. Affiliated to a social security system (except state medical aid).
6. Females: At the time of enrollment, negative human chorionic gonadotropin (hCG) pregnancy test (serum) for women presumed to be of childbearing potential on the day of enrollment. On Day 1 (pre-vaccination): negative urine pregnancy test (hCG), (only required if serum pregnancy test was performed more than 3 days before).

   Note: Women that are postmenopausal (defined as amenorrhea for ≥ 12 consecutive months prior to screening [Day 1]) or permanently sterilized will be considered as not having reproductive potential.
7. Females of childbearing potential must use highly effective of birth control from 1 month before the first administration of the trial vaccine until 3 months following the last administration. The following methods of birth control are considered highly effective when used consistently and correctly:

   * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal);
   * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable);
   * Intrauterine devices (IUDs);
   * Intrauterine hormone-releasing systems (IUSs);
   * Bilateral tubal occlusion;
   * Vasectomized partner.
   * Same sex relationships.

Sexual abstinence (periodic abstinence [e.g., calendar, ovulation symptothermal and post-ovulation methods]) and withdrawal are not acceptable methods.

Exclusion Criteria:

1. Participant ill or febrile (body temperature ≥38.0°C) within 72 hours prior to screening and/or symptoms suggestive of coronavirus disease 2019 (COVID-19) within the past 14 days prior to screening (ill or febrile participants may be re-scheduled within the predefined interval when no longer presenting symptoms).
2. Previous or currently active SARS-CoV-2 infection (currently as confirmed by reactive polymerase chain reaction [PCR] or positive serology test prior to the first trial vaccine administration).
3. Use of any investigational or non-registered product (vaccine or drug) other than the trial vaccine within 28 days preceding the administration of the trial vaccine, or planned use during the trial period.
4. Receipt of any other vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrollment in this trial or planned receipt of any vaccine within 28 days of trial vaccine administration.
5. Receipt of any investigational or licensed/authorized SARS-CoV-2 or other coronavirus vaccine, including non-specific vaccines such as Bacillus Calmette-Guérin, prior to the administration of the trial vaccine or planned administration during the trial.
6. Any treatment with immunosuppressants or other immune-modifying drugs (including, but not limited to, corticosteroids, biologicals and Methotrexate) for > 14 days total within 6 months preceding the administration of trial vaccine or planned use during the trial. For corticosteroid use, this means prednisone or equivalent, 0.5 mg/kg/day for 14 days or more. The use of inhaled, topical, or localized injections of corticosteroids (e.g., for joint pain/inflammation) is permitted.
7. Receipt of any lipid nanoparticles (LNP)-formulated messenger ribonucleic acid vaccine prior to the administration of the trial vaccine.
8. Any medically diagnosed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination, including known human immunodeficiency virus infection, hepatitis B virus infection and hepatitis C virus infection.
9. History of potential immune-mediated disease.
10. History of angioedema.
11. Any known allergy to any component of investigational CVnCoV or aminoglycoside antibiotics.
12. History of or current alcohol and/or drug abuse.
13. History of severe acute respiratory syndrome (SARS) or Middle East respiratory syndrome (self-reported).
14. Administration of immunoglobulins (Igs) and/or any blood products within the 3 months preceding the administration of any dose of the trial vaccine or planned administration during the trial.
15. Participants with a significant acute or chronic medical or psychiatric illness that, in the opinion of the Investigator, precludes trial participation (e.g., may increase the risk of trial participation, render the participant unable to meet the requirements of the trial, or may interfere with the participant's trial evaluations). These include severe and/or uncontrolled cardiovascular disease, gastrointestinal disease, liver disease, renal disease, respiratory disease, endocrine disorder, and neurological and psychiatric illnesses. However, those with controlled and stable cases can be included in the trial.
16. Foreseeable non-compliance with protocol as judged by the Investigator.
17. For females: pregnancy or lactation.
18. History of any anaphylactic reactions.
19. Participants with a significant bleeding disorder (e.g., factor deficiency, coagulopathy or platelet disorder) or prior history of significant bleeding or bruising following intramuscular (IM) injections or venipuncture.
20. Participants employed by the Sponsor, Investigator or trial site, or relatives of research staff working on this trial.
21. Participant is committed to an institution (by virtue of an order issued either by the judicial or the administrative authorities).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Antibody Concentrations Against SARS-CoV-2 Spike Protein-specific Immunoglobulin G (IgG) in Serum | Day 43
  Measured by enzyme-linked immunosorbent assay (ELISA).

SECONDARY OUTCOMES:
Antibody Concentrations Against SARS-CoV-2 Spike Protein-specific Immunoglobulin G (IgG) in Serum | Month 6, Month 12 and Month 26
  Measured by enzyme-linked immunosorbent assay (ELISA).
Antibody Concentrations Against SARS-CoV-2 Spike Protein-specific Immunoglobulins in Serum | Day 29, Day 43, Month 6, Month 12 and Month 26
  Antibody concentrations against SARS-CoV-2 spike protein-specific immunoglobulin A (IgA) and immunoglobulin M (IgM) in serum.
  Measured by enzyme-linked immunosorbent assay (ELISA).
Number of Participants With Neutralizing Antibody Titers Against SARS-CoV-2 Spike Protein in Serum | Day 29, Day 43, Month 6, Month 12 and Month 26
  Measured by an in vitro neutralization assay.
Number of Participants Who Experience a Solicited Local Adverse Event (AE) | Up to 7 days after vaccination
Intensity of Solicited Local Adverse Events (AEs) per the US Food and Drug Administration (FDA) Toxicity Grading Scale | Up to 7 days after vaccination
  Intensity of solicited local AEs will be graded per the FDA Toxicity Grading Scale at grades 0-3, where higher grades indicate a worse outcome.
Duration of Solicited Local Adverse Events (AEs) | Up to 7 days after vaccination
Number of Participants Who Experience a Solicited Systemic Adverse Event (AE) | Up to 7 days after vaccination
Intensity of Solicited Systemic Adverse Events (AEs) per the US Food and Drug Administration (FDA) Toxicity Grading Scale | Up to 7 days after vaccination
  Intensity of solicited systemic AEs will be graded per the FDA Toxicity Grading Scale at grades 0-3, where higher grades indicate a worse outcome.
Duration of Solicited Systemic Adverse Events (AEs) | Up to 7 days after vaccination
Number of Participants Who Experience a Treatment-related Solicited Systemic Adverse Event (AE) | Up to 7 days after vaccination
Number of Participants Who Experience an Unsolicited Adverse Event (AE) | Up to 28 days after vaccination
Intensity of Unsolicited Adverse Events (AEs) per the Investigator's Assessment | Up to 28 days after vaccination
Number of Participants Who Experience a Treatment-related Unsolicited Adverse Event (AE) | Up to 28 days after vaccination
Number of Participants Who Experience a Medically Attended Adverse Event (AE) | Day 1 up to approximately 26 months
Number of Participants Who Experience a Treatment-related Medically Attended Adverse Event (AE) | Day 1 up to approximately 26 months
Number of Participants Who Experience a Medically Attended Serious Adverse Event (SAE) | Day 1 up to approximately 26 months
Number of Participants Who Experience a Medically Attended Treatment-related Serious Adverse Event (SAE) | Day 1 up to approximately 26 months
Number of Participants Who Experience a Medically Attended Adverse Event of Special Interest (AESI) | Day 1 up to approximately 26 months
Number of Participants Who Experience a Treatment-related Medically Attended Adverse Event of Special Interest (AESI) | Day 1 up to approximately 26 months
Number of Participants With Virologically-confirmed SARS-CoV-2 Infection | Screening up to approximately 26 months
  Measured by reverse transcription polymerase chain reaction (RT-PCR).